CLINICAL TRIAL: NCT00010686
Title: Dietary Phytoestrogens and Bone Metabolism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: P50AT000090-01P2 (NIH); P50AT000090-01 (NIH); NCT00009360 (obsolete NCT alias)
Record Dates: First submitted 2001-02-02; First posted 2001-02-05 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2006-08

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis

INTERVENTIONS:
Drug: Dietary Phytoestrogens

SUMMARY:
The purpose of this study is to determine whether dietary phytoestrogens are an effective alternative to postmenopausal exogenous estrogen replacement therapy in preventing bone loss.

DETAILED DESCRIPTION:
Osteoporosis in postmenopausal women is one of the most important public health challenges of our time. With millions of women affected and billions of dollars being spent for its complications, we need to develop effective approaches to this disease. Postmenopausal women are at particular risk because the loss of estrogen associated with the menopause leads to bone loss of much greater magnitude than one would expect on the basis of age alone. Estrogen replacement therapy, a logical and effective therapeutic approach, has been associated with serious concerns about adverse events and, thus, limited use. The recent development of selective estrogen receptor modulators (SERMS) may help if they continue to show promise. Interest in natural sources of estrogenic substances to prevent postmenopausal bone loss is an expected outgrowth of the general interest in alternative medicinals for a wide variety of human disorders. Concerns about the potential for adverse consequences of the conventional use of estrogen replacement therapy, and limited knowledge about long term use of SERMS- add support to this quest. No systematic investigation of the role of dietary phytoestrogens on bone mass and skeletal dynamics has yet been conducted. With the dramatic increase in interest in these sources of estrogenic activity, it is important for us to determine whether these agents are efficacious. Otherwise, this field will be plagued for years to come by incomplete, anecdotal and scientifically poorly documented actions of these agents on bone metabolism. It is our expectation that this study will begin to provide the documentary information that the field so clearly needs. The rationale for exploring the potential for phytoestrogens in the maintenance of skeletal health in postmenopausal women is clear and compelling.

Women will be randomly assigned to one of three healthy eating plans and, over the course of the year-long study, will learn to choose and cook foods to help optimize health as they go through menopause and beyond.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal
* Weight within 90% to 120% of ideal body weight
* 12 or more months since last menstrual period
* New York Metro Area resident

Exclusion Criteria:

* History of cancer, diabetes, or heart disease
* Smoker

Ages: 50 Years to 72 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Study Completion 2005-12

CONTACTS AND LOCATIONS:
Overall Officials: Dr. John P. Bilezikian, Principal Investigator — Columbia University
Locations (1):
- Columbia University/Health Science Division, New York, New York, United States